CLINICAL TRIAL: NCT01504399
Title: Rhinological Outcomes in Endonasal Pituitary Surgery: A Multi-Center Observational Cohort Study
Brief Title: Rhinological Outcomes in Endonasal Pituitary Surgery
Status: Completed | Type: Observational
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Responsible Party: Sponsor
Other Study IDs: 11BN093
Record Dates: First submitted 2012-01-03; First posted 2012-01-05 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Pituitary Neoplasm; Pituitary Adenoma; Prolactinoma; Cushings Disease; Acromegaly
Keywords: Pituitary surgery; Transsphenoidal surgery; Anterior skull base surgery; Endoscopic surgery; Patient survey; Nasal complications
MeSH Terms: conditions — Pituitary Neoplasms; Prolactinoma; Adrenocortical Hyperfunction; Acromegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Microscopic:: Microscopic (single nostril, direct endonasal with nasal speculum)transsphenoidal nasal surgery
- Endoscopic: Fully endoscopic: (bi-nostril, no nasal speculum) transsphenoidal pituitary surgery

SUMMARY:
This is a prospective, multi-center observational study designed to address patient-reported nasal outcomes in adults undergoing endoscopic and microscopic surgical removal of pituitary tumors. The primary objective of this study is to determine the difference in nasal outcomes by using the Anterior Skull Base (ASK) Nasal survey between patients treated with endoscopic surgical technique and those treated with microscopic surgical technique. Patients will be given the ASK Nasal survey to assess their nasal functioning and overall health before their surgery, and at post-operative visits 1-2 weeks, 3 months, and 6 months.

DETAILED DESCRIPTION:
The technical and patient factors that influence rhinological (nasal) outcomes following endonasal anterior skull base surgery and pituitary surgery are not well understood. Several timely and controversial topics, such as the influence of endoscopic techniques and the impact of underlying disease on nasal outcomes are in need of further study.

The Anterior Skull Base (ASK) Nasal survey is a 24-item questionnaire designed to assess for common postoperative nasal complaints, such as crusting, nasal congestion, pain, sinusitis, sense of smell, and overall functioning. The survey is a brief and simple assessment that asks patients to score symptom severity on a five-point scale.

ELIGIBILITY:
Inclusion Criteria:

* Pituitary tumor patients treated by transsphenoidal route
* Adults (age 18-80 years)
* Direct endonasal or endoscopic approach
* Non-functioning adenoma, Cushing's disease, acromegaly

Exclusion Criteria:

* Patients treated by expanded endonasal approaches (transtubercular approach)
* Sublabial approach

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pituitary lesions referred to our investigators for surgical management by either microscopic or endoscopic transspenoidal surgical resection.
Sampling Method: Non-Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2011-10-01 (Actual); Primary Completion 2014-06-01 (Actual); Study Completion 2015-12-09 (Actual)

PRIMARY OUTCOMES:
ASK Nasal symptom severity scores and SF-8 scores | 3 months
  Compare symptom severity scores and quality of life scores in first-time surgery patients with nonfunctioning adenomas on the ASK Nasal and SF-8.
Validation of ASK Nasal survey tool | 3 months
  Validate a nasal outcomes scale (ASK Nasal) specifically designed for anterior skull base surgery.

SECONDARY OUTCOMES:
ASK Nasal symptom severity scores | 2 weeks, 3 months, 6 months postoperative
  * Evaluate the symptom severity scores on the ASK Nasal for first time surgery patients with nonfuctioning adenomas at the first post-operative visit and at 6 months.
  * Evaluate the symptom severity scores on the ASK Nasal for all patients at the first post-operative visit and at 6 months.
Impact of surgical techniques and complications on ASK Nasal scores | 6 months
  * Subgroup analysis on the impact of such surgical techniques, such as middle turbinate resection and nasal packing, on ASK Nasal scores will be performed.
  * Subgroup analysis of rhinological complications, such as sinusitis, on ASK Nasal scores.
  * Objective intranasal endoscopy findings at follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S. Little, MD, Principal Investigator — Barrow Neurological Institute at St. Joseph's Hospital and Medical Center
Locations (4):
- United States (4):
  - Barrow Neurological Institute/St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - John Wayne Cancer Institute at St. John's Health Center, Santa Monica, California
  - Northshore University Health System, Chicago, Illinois
  - Ohio State University Medical Center, Columbus, Ohio

REFERENCES:
- [Background] Little AS, Jahnke H, Nakaji P, Milligan J, Chapple K, White WL. The anterior skull base nasal inventory (ASK nasal inventory): a clinical tool for evaluating rhinological outcomes after endonasal surgery for pituitary and cranial base lesions. Pituitary. 2012 Dec;15(4):513-7. doi: 10.1007/s11102-011-0358-4. PMID 22038032
- [Derived] Zaidi HA, Awad AW, Bohl MA, Chapple K, Knecht L, Jahnke H, White WL, Little AS. Comparison of outcomes between a less experienced surgeon using a fully endoscopic technique and a very experienced surgeon using a microscopic transsphenoidal technique for pituitary adenoma. J Neurosurg. 2016 Mar;124(3):596-604. doi: 10.3171/2015.4.JNS15102. Epub 2015 Oct 16. PMID 26473774
- [Derived] Little AS, Kelly DF, Milligan J, Griffiths C, Prevedello DM, Carrau RL, Rosseau G, Barkhoudarian G, Jahnke H, Chaloner C, Jelinek KL, Chapple K, White WL. Comparison of sinonasal quality of life and health status in patients undergoing microscopic and endoscopic transsphenoidal surgery for pituitary lesions: a prospective cohort study. J Neurosurg. 2015 Sep;123(3):799-807. doi: 10.3171/2014.10.JNS14921. Epub 2015 Apr 17. PMID 25884256
- [Derived] Little AS, Kelly D, Milligan J, Griffiths C, Prevedello DM, Carrau RL, Rosseau G, Barkhoudarian G, Otto BA, Jahnke H, Chaloner C, Jelinek KL, Chapple K, White WL. Predictors of sinonasal quality of life and nasal morbidity after fully endoscopic transsphenoidal surgery. J Neurosurg. 2015 Jun;122(6):1458-65. doi: 10.3171/2014.10.JNS141624. Epub 2015 Apr 3. PMID 25839931
- [Derived] Little AS, Kelly D, Milligan J, Griffiths C, Rosseau G, Prevedello DM, Carrau R, Jahnke H, Chaloner C, O'Leary J, Chapple K, Nakaji P, White WL. Prospective validation of a patient-reported nasal quality-of-life tool for endonasal skull base surgery: The Anterior Skull Base Nasal Inventory-12. J Neurosurg. 2013 Oct;119(4):1068-74. doi: 10.3171/2013.3.JNS122032. Epub 2013 May 10. PMID 23662829